CLINICAL TRIAL: NCT07289126
Title: Sonographic Evaluation of Ovarian Masses by ORADS System in Woman's Health Hospital
Brief Title: Sonographic Evaluation of Ovarian Masses by ORADS System
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Emad Eldin Mostafa, Resident at Obstetrics and Gynecology Department, Assiut University, Assiut University
Other Study IDs: evaluation of ovarian masses
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sonography; Ovarian Mass
Keywords: ovarian masses; ORADS system; Ovarian-Adnexal Reporting and Data System Ultrasound; sonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Benign Ovarian Masses: Women aged 18-70 years with ovarian cysts or masses detected on transabdominal or transvaginal ultrasound, whose lesions are finally confirmed as benign by histopathology after standard clinical management, including ultrasound evaluation by O-RADS, MRI (when indicated), and surgical exploration or follow-up.
- Malignant Ovarian Masses: Women aged 18-70 years with ovarian cysts or masses detected on transabdominal or transvaginal ultrasound, whose lesions are finally confirmed as malignant by histopathology after standard clinical management, including ultrasound evaluation by O-RADS, MRI (when indicated), and surgical exploration.

SUMMARY:
This observational study will evaluate how well an ultrasound scoring system called O-RADS can distinguish between benign (non-cancerous) and malignant (cancerous) ovarian masses in women aged 18 to 70 years. Women who are found to have an ovarian cyst or mass during routine pelvic or transabdominal ultrasound at Women's Health Hospital will be invited to participate and will receive standard care, including detailed transvaginal ultrasound, MRI when indicated, surgery if needed, and histopathology (tissue examination). The main question is how accurately O-RADS ultrasound categories predict the final tissue diagnosis; the study will also look at how ultrasound findings relate to MRI results in characterizing ovarian masses.

DETAILED DESCRIPTION:
This is a prospective cross-sectional diagnostic accuracy study designed to evaluate the performance of the Ovarian-Adnexal Reporting and Data System (O-RADS) ultrasound score in characterizing ovarian masses in women attending Woman's Health Hospital, Assiut University. The study addresses the challenge of differentiating benign from malignant adnexal lesions, a distinction that is essential for selecting appropriate management, avoiding unnecessary surgery, and optimizing referral to gynecologic oncology services.

After obtaining informed consent, eligible women with an adnexal mass detected on routine gynecologic assessment undergo standardized clinical evaluation, laboratory testing as indicated, and dedicated pelvic ultrasound, preferably transvaginal. The ultrasound examination follows the O-RADS lexicon, documenting lesion morphology (e.g., size, internal architecture, presence of solid components or papillary projections, wall/septal features, echogenicity) and Doppler vascular characteristics, and assigning an O-RADS category (0-5) reflecting estimated malignancy risk. When clinically appropriate, pelvic MRI is performed to further assess lesion characteristics. Surgical management (laparoscopy or laparotomy) is undertaken according to routine care, and histopathologic evaluation of excised tissue serves as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Any female patient with ovarian cyst or mass during routine trans-abdominal or pelvic US
* Age between 18 and 70 years.

Exclusion Criteria:

* Refusal of patients to filling consent.
* Patient with a previous history of the operated ovarian lesion
* Patient missed during follow-up or not provided pathology report.
* Pregnancy.
* Patients with functional ovarian masses ( e.g functional cysts )

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women aged 18 to 70 years attending the Women's Health Hospital, Assiut University, with ovarian cysts or masses detected on routine transabdominal or transvaginal ultrasound will be invited to participate. Eligible patients will undergo standardized clinical assessment, ultrasound evaluation using the O-RADS system, MRI when clinically indicated, and subsequent surgical exploration and histopathological examination or follow-up according to usual care. Patients with prior ovarian surgery for the same lesion, pregnancy, functional ovarian cysts, or those who decline consent or are lost before histopathological confirmation will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of O-RADS ultrasound in differentiating benign from malignant ovarian masses | From initial ultrasound examination to availability of final histopathology report for each participant (estimated up to 3 months).
  Proportion of correctly classified ovarian masses using the O-RADS ultrasound scoring system compared with the reference standard of postoperative histopathological diagnosis (benign vs malignant). Accuracy will be expressed as sensitivity, specificity, positive predictive value, negative predictive value, and overall accuracy for O-RADS categories indicating malignancy.